CLINICAL TRIAL: NCT03741543
Title: Learning and Coping With Dementia - User Experiences From an Educative Intervention in Early Stage Dementia
Brief Title: Learning and Coping With Early Stage Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: The Dam Foundation (Other); The National Association for Public Health, Norway (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: sus2018mk01
Record Dates: First submitted 2018-11-06; First posted 2018-11-15 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Dementia; Alzheimer Disease; Vascular Dementia
Keywords: health promotion; early-stage dementia; psychosocial
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular | interventions — Psychosocial Intervention

STUDY DESIGN:
Intervention Model Description: a 12-week health promotion course
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A 12-week health promotion course (Other): The Health Promotion intervention consists of 12 weekly 2-hour sessions with a group of up to six participants and two course facilitators. Teaching methods includes lecture, questions- and answer periods, and interactive hands-on learning. During the class sessions, the facilitators encourages the participants to ask questions and make comments about the lecture at any time. During the first class session, each participant receives a booklet with the course material
  Interventions: Other: A 12-week health promotion course

INTERVENTIONS:
Other: A 12-week health promotion course — The Health Promotion intervention consists of 12 weekly 2-hour sessions with a group of up to six participants and two course facilitators. Teaching methods includes lecture, questions- and answer periods, and interactive hands-on learning. During the class sessions, the facilitators encourages the participants to ask questions and make comments about the lecture at any time. During the first class session, each participant receives a booklet with the course material.
  Other Names: Psychosocial intervention, group based

SUMMARY:
The overall aim of this study is to investigate how home dwelling people with early-stage dementia cope with their disease, explored through their participation in a 12-week health promotion course, through 3 sub-studies; 1) The users' experience in gaining information about dementia and meeting others in the same situation, 2) observation of the group interactions and support processes, and 3) investigate the effect of the 12-week health promotion course for people with early stage dementia on their cognitive function, psychosocial function and health behaviour.

DETAILED DESCRIPTION:
In this study, the investigators build on a health promotion intervention originally developed by Buettner and Fitzimmons (2009), called "Health Promotion for the Mind, Body, and Spirit". The Health Promotion intervention consists of 12 weekly 2-hour sessions. Each group has up to 6 participants, and the groups are facilitated by two professional group leaders. The course has been designed to provide information on the disease process and on healthy behaviours to prevent problems that are common later in the disease. The 12-week course includes nutrition, cognitive fitness, stress reduction, communication, information about the course of the disease, and coping strategies. During the first class session, each participant received a nametag and a booklet. This booklet is a critical component of the educational method for the participants. The booklet contains 12 dividers for the 12 modules that the instructor taught during the course. The caregiver is not present at the course, however the participants are encouraged to share the booklet provided at the course with the caregiver between sessions.

Design: a quasi-experimental study with multiple methods:

1. assessment of cognitive function, psychosocial function and health behaviour is collected at baseline (prior to attending the 12-week course) and follow-up interviews are arranged shortly after the 12-week course. For each participant a caregiver also has to take part for proxy interviews.
2. the users' experience of attending the 12-week health promotion course will be collected through qualitative individual interviews with the participants and their caregiver after attending the course.
3. over the duration of the course a moderate participant observation will be carried out to explore changes over the 12-week course, in-session behaviour, social interaction and to capture motivational and empowering aspects of the course.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* A diagnosis of early or moderate stage dementia
* Capable of reading and writing
* Hearing and vision which are sufficiently good to work in a group setting
* Proficient in the language in which the course is provided

Exclusion Criteria:

* A diagnosis of alcohol abuse
* A limited life expectancy due to any terminal disease or other serious illness
* Chemotherapy or radiation treatment ongoing at enrolment
* Head injuries
* Epilepsy
* Parkinson's disease
* A history of psychiatric illness
* A history of a diagnosis of subnormal intelligence
* Prior participation in health promotion or cognitive training programs

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The users experiences from an educative intervention in early-stage dementia | Baseline, 3 months
  Qualitative data will be collected through semi-structured individual interviews with both participants and their caregiver (proxy), and through moderate participant observations following the participants over the duration of the 12-week course. The interview guide and observational protocol consist of pre-selected topics, including (1) communication, (2) participant engagement, (3) social interaction within the group, (4) peer support (5) change in perception of living with dementia and (6) educational outcome. The qualitative data will be explored using content analysis.

SECONDARY OUTCOMES:
Change in cognitive function | Baseline, 3 months
  Measured by The Mini Mental State Examination (MMSE)
Change in depressive symptoms | Baseline, 3 months
  Depressive symptoms will be measured by the Cornell Scale for Depression in Dementia (CSDD) (Alexopoulos et al., 1988).The CSDD is an assessment of signs and symptoms of depression in people with dementia. Each item is rated for severity on a scale of 0-2 (0=absent, 1=mild or intermittent, 2=severe). Sum score above 10 indicate a probable major depression. Scores above 18 indicate a definite major depression. Scores below 6 are associated with absence of significant depressive symptoms.
Change in self-rated health | Baseline, 3 months
  Self-rated health will be measured by The EuroQol visual analogue scale (VAS) (The EuroQol group, 1990). The EQ VAS measures the participants self-rated Health-Related Quality of Life on a vertical, visual analogue scale, form 0-100. Where 0 presents "worst imaginable health state" and 100 represents "best-imagined health state".
Change in managing personal activities of daily life | Baseline, 3 months
  The levels of personal functioning in daily life will be measured by Lawton and Brody's Physical Self-Maintenance Scale. The sum-score is based on six items (range 0-30), with higher scores indicating a lower function.
Change in managing instrumental activities of daily life | Baseline, 3 months
  The levels of instrumental functioning in daily life will be measured by Instrumental Activities of Daily Living Scale (I-ADL) (Lawton et al, 1969). The I-ADL sum-score is based on eight items (range 0-31), with higher scores indicating a lower function.
Change in neuropsychiatric symptoms | Baseline, 3 months
  Neuropsychiatric symptoms will be assessed using The Neuropsychiatric Inventory (NPI) (Cummings, et al., 1994), a 12-item questionnaire developed to assess behavioural disturbances in people with dementia. Scores are entered for the frequency and degree of seriousness of each symptom over the last four weeks, and subsequently multiplied into a symptom score. The total possible maximum score is 144. A higher score reflects increased frequency and severity of the disturbances.
Change in carer stress/burden | Baseline, 3 months
  To measure caregiver burden the Relative Stress Scale (RSS), will be used. RSS assesses the caregiver burden for people caring for individuals with dementia. The RSS has 15 different questions, each scored 0-4 (0=never/not at all, 1=rarely/a little, =sometimes/moderately, 3=frequently/quite a lot, 4=always/considerably perceived burden), with a total score range of 0-60. Higher scores reflect a higher reported caregiver burden.

CONTACTS AND LOCATIONS:
Overall Officials: Ingelin Testad, PhD, Principal Investigator — Helse Stavanger

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buettner LL, Fitzsimmons S. Promoting health in early-stage dementia: evaluation of a 12-week course. J Gerontol Nurs. 2009 Mar;35(3):39-49. doi: 10.3928/00989134-20090301-02. PMID 19326828
- [Background] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Result] Testad I, Kajander M, Gjestsen MT, Dalen I. Health promotion intervention for people with early-stage dementia: A quasi-experimental study. Brain Behav. 2020 Dec;10(12):e01888. doi: 10.1002/brb3.1888. Epub 2020 Oct 16. PMID 33064358
- [Result] Kajander, M., Gjestsen, M. T., Vagle, V., Meling, M., Henriksen, A. T., & Testad, I. (2022). Health promotion in early-stage dementia-user experiences from an educative intervention. Educational Gerontology, 48(9), 391-403.
- [Result] Kajander M, Gjestsen MT, Ballard C, Naess H, Testad I. Health Promotion in Early-Stage Dementia: A Focused Ethnographic Study of a 12-Week Group-Based Educational Intervention. SAGE Open Nurs. 2024 Jul 25;10:23779608241266686. doi: 10.1177/23779608241266686. eCollection 2024 Jan-Dec. PMID 39070007
- [Result] Kajander M, Gjestsen M T, Ballard C, Naess H, Tovar-Rios D A, Fossey J, Testad I. Health promotion in early-stage dementia: Exploring associations between sociodemographic characteristics and outcomes of a 12-week group-based educational intervention. Educational Gerontology. 2024; 1-14. doi: https://doi.org/10.1080/03601277.2024.2358620

DOCUMENTS (1):
  • Study Protocol (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT03741543/Prot_000.pdf